CLINICAL TRIAL: NCT01720810
Title: Pacific Northwest Udall Center (PANUC) Clinical Core
Acronym: PANUC
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cyrus Zabetian, Professor of Neurology, University of Washington
Other Study IDs: STUDY00005005
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma, serum, CSF, brain tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study evaluates cognitive impairment in subjects with Parkinson disease (PD) and similar neurological disorder through obtaining longitudinal clinical and neuropsychological data. The long term goal is to have a well-characterized subject population to contribute to our understanding of the natural history, diagnosis and ultimate treatment of cognitive impairment in patients with PD and similar disorders.

DETAILED DESCRIPTION:
The Pacific Northwest Udall Center (PANUC) Clinical Core has recruited and characterized a cohort of more than 600 individuals with Parkinson's disease (PD) during the initial funding period. Data from the PANUC Clinical Core, in collaboration with other Udall Centers and other academic medical centers, have helped confirm apolipoprotein E (APOE) (1) and glucocerebrosidase (glucosidase, beta, acid or GBA) (2)as genes that increase the risk and modify the phenotype (1) of cognitive decline in PD. Understanding the mechanisms underlying these gene effects is the focus of this renewal application, and the Clinical Core will provide well-characterized PD and control subjects of appropriate genotypes for PANUC projects. In addition, the majority of the existing cohort will be retained for additional longitudinal clinical and neuropsychological testing follow-up to support ongoing genetic and biomarker studies, with a refined battery of tests and a uniform biannual frequency of visits designed to maximize efficiency. Balance and gait testing (already piloted at the Portland site) will be added to the test battery for the entire cohort as an innovation that is thought to reflect higher order CNS function closely related to cognition. This innovation leverages the expertise of Dr. Horak, an investigator introduced to the PANUC by way of PANUC Pilot Award funding during the last funding period. As in the current cycle, Clinical Core subjects will be followed in identical fashion at two sites: one at UW directed by Dr. Hu, and the other at OHSU directed by Core Leader Dr. Quinn. Project 3 leader Dr. Horak will oversee balance and gait testing at OHSU and Dr. Kelly will oversee balance and gait testing at UW.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson disease
* Over 18 years of age

Exclusion Criteria:

- Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects undergo the following procedures:
  * Interview to collect data on medical history and demographics
  * Neurological examination
  * Questionnaires about mood, activities of daily living, and environmental exposures.
  * Psychometric tests
  Study companions might also be asked to complete questionnaires about the participant's thinking and memory, activities of daily living, sleep, and neuropsychiatric symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Shi M, Kovac A, Korff A, Cook TJ, Ginghina C, Bullock KM, Yang L, Stewart T, Zheng D, Aro P, Atik A, Kerr KF, Zabetian CP, Peskind ER, Hu SC, Quinn JF, Galasko DR, Montine TJ, Banks WA, Zhang J. CNS tau efflux via exosomes is likely increased in Parkinson's disease but not in Alzheimer's disease. Alzheimers Dement. 2016 Nov;12(11):1125-1131. doi: 10.1016/j.jalz.2016.04.003. Epub 2016 May 24. PMID 27234211
- [Result] Morris R, Martini DN, Kelly VE, Smulders K, Ramsey K, Hiller A, Chung KA, Hu SC, Zabetian CP, Poston KL, Mata IF, Edwards KL, Lapidus J, Cholerton B, Montine TJ, Quinn JF, Horak F. Gait and balance in apolipoprotein E4 allele carriers in older adults and Parkinson's disease. Clin Park Relat Disord. 2023 May 17;9:100201. doi: 10.1016/j.prdoa.2023.100201. eCollection 2023. PMID 37252677
- [Result] Morris R, Martini DN, Ramsey K, Kelly VE, Smulders K, Hiller A, Chung KA, Hu SC, Zabetian CP, Poston KL, Mata IF, Edwards KL, Lapidus J, Cholerton B, Montine TJ, Quinn JF, Horak F. Cognition as a mediator for gait and balance impairments in GBA-related Parkinson's disease. NPJ Parkinsons Dis. 2022 Jun 20;8(1):78. doi: 10.1038/s41531-022-00344-5. PMID 35725575
- [Result] Hwangbo N, Zhang X, Raftery D, Gu H, Hu SC, Montine TJ, Quinn JF, Chung KA, Hiller AL, Wang D, Fei Q, Bettcher L, Zabetian CP, Peskind ER, Li G, Promislow DEL, Davis MY, Franks A. Predictive Modeling of Alzheimer's and Parkinson's Disease Using Metabolomic and Lipidomic Profiles from Cerebrospinal Fluid. Metabolites. 2022 Mar 22;12(4):277. doi: 10.3390/metabo12040277. PMID 35448464
- [Result] Hwangbo N, Zhang X, Raftery D, Gu H, Hu SC, Montine TJ, Quinn JF, Chung KA, Hiller AL, Wang D, Fei Q, Bettcher L, Zabetian CP, Peskind E, Li G, Promislow DEL, Franks A. A Metabolomic Aging Clock Using Human Cerebrospinal Fluid. J Gerontol A Biol Sci Med Sci. 2022 Apr 1;77(4):744-754. doi: 10.1093/gerona/glab212. PMID 34382643
- [Result] Cholerton BA, Poston KL, Yang L, Rosenthal LS, Dawson TM, Pantelyat A, Edwards KL, Tian L, Quinn JF, Chung KA, Hiller AL, Hu SC, Montine TJ, Zabetian CP. Semantic fluency and processing speed are reduced in non-cognitively impaired participants with Parkinson's disease. J Clin Exp Neuropsychol. 2021 Jul;43(5):469-480. doi: 10.1080/13803395.2021.1927995. Epub 2021 Aug 6. PMID 34355669
- [Result] Hong Z, Tian C, Stewart T, Aro P, Soltys D, Bercow M, Sheng L, Borden K, Khrisat T, Pan C, Zabetian CP, Peskind ER, Quinn JF, Montine TJ, Aasly J, Shi M, Zhang J. Development of a Sensitive Diagnostic Assay for Parkinson Disease Quantifying alpha-Synuclein-Containing Extracellular Vesicles. Neurology. 2021 May 4;96(18):e2332-e2345. doi: 10.1212/WNL.0000000000011853. Epub 2021 Mar 23. PMID 34032594
- [Result] Palmer WC, Cholerton BA, Zabetian CP, Montine TJ, Grabowski TJ, Rane S. Resting-State Cerebello-Cortical Dysfunction in Parkinson's Disease. Front Neurol. 2021 Jan 28;11:594213. doi: 10.3389/fneur.2020.594213. eCollection 2020. PMID 33584497
- [Result] Martini DN, Morris R, Madhyastha TM, Grabowski TJ, Oakley J, Hu SC, Zabetian CP, Edwards KL, Hiller A, Chung K, Ramsey K, Lapidus JA, Cholerton B, Montine TJ, Quinn JF, Horak FB. Relationships Between Sensorimotor Inhibition and Mobility in Older Adults With and Without Parkinson's Disease. J Gerontol A Biol Sci Med Sci. 2021 Mar 31;76(4):630-637. doi: 10.1093/gerona/glaa300. PMID 33252618
- [Result] Martini DN, Morris R, Kelly VE, Hiller A, Chung KA, Hu SC, Zabetian CP, Oakley J, Poston K, Mata IF, Edwards KL, Lapidus JA, Grabowski TJ, Montine TJ, Quinn JF, Horak F. Sensorimotor Inhibition and Mobility in Genetic Subgroups of Parkinson's Disease. Front Neurol. 2020 Sep 4;11:893. doi: 10.3389/fneur.2020.00893. eCollection 2020. PMID 33013627
- [Result] Rane S, Owen J, Hippe DS, Cholerton B, Zabetian CP, Montine T, Grabowski TJ. White Matter Lesions in Mild Cognitive Impairment and Idiopathic Parkinson's Disease: Multimodal Advanced MRI and Cognitive Associations. J Neuroimaging. 2020 Nov;30(6):843-850. doi: 10.1111/jon.12778. Epub 2020 Sep 16. PMID 32937003
- [Result] Phongpreecha T, Cholerton B, Mata IF, Zabetian CP, Poston KL, Aghaeepour N, Tian L, Quinn JF, Chung KA, Hiller AL, Hu SC, Edwards KL, Montine TJ. Multivariate prediction of dementia in Parkinson's disease. NPJ Parkinsons Dis. 2020 Aug 25;6:20. doi: 10.1038/s41531-020-00121-2. eCollection 2020. PMID 32885039
- [Result] Gryc W, Roberts KA, Zabetian CP, Weintraub D, Trojanowski JQ, Quinn JF, Hiller AL, Chung KA, Poston KL, Yang L, Hu SC, Edwards KL, Montine TJ, Cholerton BA. Hallucinations and Development of Dementia in Parkinson's Disease. J Parkinsons Dis. 2020;10(4):1643-1648. doi: 10.3233/JPD-202116. PMID 32741842
- [Result] Rane S, Koh N, Oakley J, Caso C, Zabetian CP, Cholerton B, Montine TJ, Grabowski T. Arterial spin labeling detects perfusion patterns related to motor symptoms in Parkinson's disease. Parkinsonism Relat Disord. 2020 Jul;76:21-28. doi: 10.1016/j.parkreldis.2020.05.014. Epub 2020 May 11. PMID 32559629
- [Result] Wilson EN, Swarovski MS, Linortner P, Shahid M, Zuckerman AJ, Wang Q, Channappa D, Minhas PS, Mhatre SD, Plowey ED, Quinn JF, Zabetian CP, Tian L, Longo FM, Cholerton B, Montine TJ, Poston KL, Andreasson KI. Soluble TREM2 is elevated in Parkinson's disease subgroups with increased CSF tau. Brain. 2020 Mar 1;143(3):932-943. doi: 10.1093/brain/awaa021. PMID 32065223
- [Result] Cholerton B, Poston KL, Tian L, Quinn JF, Chung KA, Hiller AL, Hu SC, Specketer K, Montine TJ, Edwards KL, Zabetian CP. Participant and Study Partner Reported Impact of Cognition on Functional Activities in Parkinson's Disease. Mov Disord Clin Pract. 2019 Dec 14;7(1):61-69. doi: 10.1002/mdc3.12870. eCollection 2020 Jan. PMID 31970213
- [Result] Morris R, Martini DN, Smulders K, Kelly VE, Zabetian CP, Poston K, Hiller A, Chung KA, Yang L, Hu SC, Edwards KL, Cholerton B, Grabowski TJ, Montine TJ, Quinn JF, Horak F. Cognitive associations with comprehensive gait and static balance measures in Parkinson's disease. Parkinsonism Relat Disord. 2019 Dec;69:104-110. doi: 10.1016/j.parkreldis.2019.06.014. Epub 2019 Jul 4. PMID 31731260
- [Result] Specketer K, Zabetian CP, Edwards KL, Tian L, Quinn JF, Peterson-Hiller AL, Chung KA, Hu SC, Montine TJ, Cholerton BA. Visuospatial functioning is associated with sleep disturbance and hallucinations in nondemented patients with Parkinson's disease. J Clin Exp Neuropsychol. 2019 Oct;41(8):803-813. doi: 10.1080/13803395.2019.1623180. Epub 2019 Jun 10. PMID 31177941
- [Result] Hendershott TR, Zhu D, Llanes S, Zabetian CP, Quinn J, Edwards KL, Leverenz JB, Montine T, Cholerton B, Poston KL. Comparative sensitivity of the MoCA and Mattis Dementia Rating Scale-2 in Parkinson's disease. Mov Disord. 2019 Feb;34(2):285-291. doi: 10.1002/mds.27575. Epub 2018 Dec 10. PMID 30776152
- [Result] Kim HM, Nazor C, Zabetian CP, Quinn JF, Chung KA, Hiller AL, Hu SC, Leverenz JB, Montine TJ, Edwards KL, Cholerton B. Prediction of cognitive progression in Parkinson's disease using three cognitive screening measures. Clin Park Relat Disord. 2019;1:91-97. doi: 10.1016/j.prdoa.2019.08.006. Epub 2019 Oct 20. PMID 32368733
- [Result] Cholerton B, Johnson CO, Fish B, Quinn JF, Chung KA, Peterson-Hiller AL, Rosenthal LS, Dawson TM, Albert MS, Hu SC, Mata IF, Leverenz JB, Poston KL, Montine TJ, Zabetian CP, Edwards KL. Sex differences in progression to mild cognitive impairment and dementia in Parkinson's disease. Parkinsonism Relat Disord. 2018 May;50:29-36. doi: 10.1016/j.parkreldis.2018.02.007. Epub 2018 Feb 9. PMID 29478836
- [Result] Licking N, Murchison C, Cholerton B, Zabetian CP, Hu SC, Montine TJ, Peterson-Hiller AL, Chung KA, Edwards K, Leverenz JB, Quinn JF. Homocysteine and cognitive function in Parkinson's disease. Parkinsonism Relat Disord. 2017 Nov;44:1-5. doi: 10.1016/j.parkreldis.2017.08.005. Epub 2017 Aug 9. PMID 28807493
- [Result] Mata IF, Johnson CO, Leverenz JB, Weintraub D, Trojanowski JQ, Van Deerlin VM, Ritz B, Rausch R, Factor SA, Wood-Siverio C, Quinn JF, Chung KA, Peterson-Hiller AL, Espay AJ, Revilla FJ, Devoto J, Yearout D, Hu SC, Cholerton BA, Montine TJ, Edwards KL, Zabetian CP. Large-scale exploratory genetic analysis of cognitive impairment in Parkinson's disease. Neurobiol Aging. 2017 Aug;56:211.e1-211.e7. doi: 10.1016/j.neurobiolaging.2017.04.009. Epub 2017 Apr 20. PMID 28526295
- [Result] Yang L, Stewart T, Shi M, Pottiez G, Dator R, Wu R, Aro P, Schuster RJ, Ginghina C, Pan C, Gao Y, Qian W, Zabetian CP, Hu SC, Quinn JF, Zhang J. An alpha-synuclein MRM assay with diagnostic potential for Parkinson's disease and monitoring disease progression. Proteomics Clin Appl. 2017 Jul;11(7-8):10.1002/prca.201700045. doi: 10.1002/prca.201700045. Epub 2017 Apr 19. PMID 28319654
- [Result] Cooper CA, Jain N, Gallagher MD, Weintraub D, Xie SX, Berlyand Y, Espay AJ, Quinn J, Edwards KL, Montine T, Van Deerlin VM, Trojanowski J, Zabetian CP, Chen-Plotkin AS. Common variant rs356182 near SNCA defines a Parkinson's disease endophenotype. Ann Clin Transl Neurol. 2016 Nov 25;4(1):15-25. doi: 10.1002/acn3.371. eCollection 2017 Jan. PMID 28078311
- [Result] Irwin DJ, Grossman M, Weintraub D, Hurtig HI, Duda JE, Xie SX, Lee EB, Van Deerlin VM, Lopez OL, Kofler JK, Nelson PT, Jicha GA, Woltjer R, Quinn JF, Kaye J, Leverenz JB, Tsuang D, Longfellow K, Yearout D, Kukull W, Keene CD, Montine TJ, Zabetian CP, Trojanowski JQ. Neuropathological and genetic correlates of survival and dementia onset in synucleinopathies: a retrospective analysis. Lancet Neurol. 2017 Jan;16(1):55-65. doi: 10.1016/S1474-4422(16)30291-5. PMID 27979356
- [Result] Davis MY, Johnson CO, Leverenz JB, Weintraub D, Trojanowski JQ, Chen-Plotkin A, Van Deerlin VM, Quinn JF, Chung KA, Peterson-Hiller AL, Rosenthal LS, Dawson TM, Albert MS, Goldman JG, Stebbins GT, Bernard B, Wszolek ZK, Ross OA, Dickson DW, Eidelberg D, Mattis PJ, Niethammer M, Yearout D, Hu SC, Cholerton BA, Smith M, Mata IF, Montine TJ, Edwards KL, Zabetian CP. Association of GBA Mutations and the E326K Polymorphism With Motor and Cognitive Progression in Parkinson Disease. JAMA Neurol. 2016 Oct 1;73(10):1217-1224. doi: 10.1001/jamaneurol.2016.2245. PMID 27571329